CLINICAL TRIAL: NCT02915926
Title: Occupational Performance Coaching in Mothers of Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Welfare and Rehabilitation Science (Other)
Responsible Party: Principal Investigator, mina ahmadi kahjoogh, principal investigator, University of Social Welfare and Rehabilitation Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR.USWR.REC.1395.148
Record Dates: First submitted 2016-09-21; First posted 2016-09-27 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OT (Active Comparator): standard OT
  Interventions: Behavioral: standard OT
- OT+OPC (Experimental): occupational performance coaching
  Interventions: Behavioral: occupational performance coaching; Behavioral: standard OT

INTERVENTIONS:
Behavioral: occupational performance coaching
  Arms: OT+OPC
Behavioral: standard OT

SUMMARY:
A single-blind Randomized Controlled Trial will be used to test the efficacy of the OPC on self-efficacy and occupational performance with mothers of children with cerebral palsy. Canadian Occupational Performance Measurement and Sherer general self-efficacy scale will be employed to data collection. The sample size was determined for each group of 15 people. The participants conveniently and according to inclusion and exclusion criteria will be randomized into the groups. Participants in the intervention group will be participated in 10 sessions of OPC. At the end the questionnaires will be completed by both groups.

ELIGIBILITY:
Inclusion Criteria:

mothers: being literate 25 to 25 caring nobody disabled other than her child children: 5 to 12 cerebral palsy

Exclusion Criteria:

children: others problems that affect on communication

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2017-01-19 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | 10 weeks
  It is a questionnaire.

SECONDARY OUTCOMES:
Sherer general self-efficacy | 10 weeks
  It is a questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Mina Ahmadi Kahjoogh, Tehran, Iran